CLINICAL TRIAL: NCT00548301
Title: Study of Cyclosporine in the Treatment of Dry Eye Syndrome (ST-603-007)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sirion Therapeutics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: ST-603-007
Record Dates: First submitted 2007-10-22; First posted 2007-10-23 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2011-06

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cyclosporine

INTERVENTIONS:
Drug: cyclosporine

SUMMARY:
The purpose of this phase 3 study is to determine the safety and efficacy of cyclosporine in the treatment of dry eye syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate to severe dry eye syndrome with or without Sjogren's syndrome or other autoimmune disease

Exclusion Criteria:

* Intraocular or refractive surgery in the study eye within 3 months prior to study start
* Unwilling to discontinue use of contact lenses during the run-in and duration of the study
* Pregnancy or lactation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Roger Vogel, MD, Study Chair — Sirion Therapeutics
Locations (1):
- Eye Center Northeast, Bangor, Maine, United States